CLINICAL TRIAL: NCT04807933
Title: Neurovegetative Decoupling in the Visceral-brain Axis and Cognitive-emotional Vulnerability in Somatoform Disorders : Interest of Vagal Biofeedback
Brief Title: Neurovegetative Decoupling in Somatoform Disorders : Biofeedback Interest
Acronym: BIOFEESOMATO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The clinical trial is finished
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Laboratoire de Psychologie et NeuroCognition (Other); Laboratoire interuniversitaire de psychologie - LIP-PC2S (Unknown)
Responsible Party: Principal Investigator, Essaiclinique_BIOFEESOMATO, Pr. Bruno Bonaz, University Hospital, Grenoble
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2020-A02155-34
Record Dates: First submitted 2021-03-01; First posted 2021-03-19 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Somatoform Disorders; Irritable Bowel Syndrome; Psychogenic Non-Epileptic Seizure
Keywords: Autonomic nervous system; Brain-gut axis; Endophenotype; Cognitive-emotional vulnerability; Traumas; Biofeedback; Heart rate variability; Vagal tone; Central nervous system; Enteric nervous system; Early life events; Somatoform disorders; Stress; Irritable bowel syndrome; Psychogenic non epileptic seizures
MeSH Terms: conditions — Somatoform Disorders; Irritable Bowel Syndrome; Psychogenic Nonepileptic Seizures; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: The study requires 3 sessions (T1 / T2 / T3) with at least 24 days between each. The period (24 days) between the first session and the second session (T1-T2) will be considered as the control period. During the period, the participants will practice none exercise. The period (24 days) between the second session and the third session (T2-T3) will be considered as the intervention period. At the end of the second session (T2), the participants will be separated into two inter-subject groups: an experimental group performing BFB technique (3X5 min per day) in the intervention period (T2-T3) and a control group not performing a specific exercise in the intervention period (T2-T3).
Who Masked: Participant
Masking Description: The participants won't be informed of the condition to which they belong. A debriefing will be done at the end of the last session (T3) for each participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (BFB training) (Experimental): The participants assigned to the experimental group will do the biofeedback training using the Emwave software during the intervention period (T2-T3). The biofeedback software (Emwave Pro®) includes a photoplethysmography sensor that can be positioned on the earlobe. The installation of the program and the explanations needed for using it, will be done during the second session (T2). According to the guidelines, a fractional training is proposed 5 minutes, 3 times a day for 24 days (T2-T3).
  Interventions: Behavioral: Heart rate variability Biofeedback [HRV-BFB]
- Control group (no BFB training) (No Intervention): The participants assigned to the experimental group will not do a specific exercise during the intervention period (T2-T3).

INTERVENTIONS:
Behavioral: Heart rate variability Biofeedback [HRV-BFB] — BFB consists of a physiological recording used as a visual physiological feedback that can teach us how to control our physiology, which is naturally unconscious and uncontrollable. The BFB focused on the heart rate variability (HRV-BFB) could regulate the autonomic nervous system (vagal tone and sympathetic-parasympathetic balance) and the emotional state. The HRV BFB has received several clinical and experimental confirmations as a physiological remediation method. It is an innovative and non-pharmacological therapy frequently used to relieve stress.
  Other Names: Complementary technique
  Arms: Experimental group (BFB training)

SUMMARY:
Evaluation of the physiological and clinical effects of the biofeedback training with patients suffering from somatoform disorders, depending on their neurovegetative profile related to a visceral-brain decoupling.

DETAILED DESCRIPTION:
Somatoform disorders [SD] are defined as physiological function or organ disturbances unexplained by a specific diagnosis criterion. Some approaches have recently defended the idea of common factors of vulnerability behind the large variability of the clinical symptoms regarding the SD. In this context, the lead of the neurovegetative disturbances started receiving attention following some studies that suggested the autonomic nervous system [ANS] disturbances concerning a somatoform disorder, independently of its form. Two different neurovegetative endophenotypes (individual autonomic profiles) were highlighted: a functional neurovegetative profile (high vagal tone) and a dysfunctional neurovegetative profile (low vagal tone).

A dysfunctional neurovegetative profile could be accompanied by a chronic decoupling in the brain-visceral axis according as the ANS is considered as a bidirectional communication system linked the central nervous system [CNS] and the viscera. Depending on the types of the neurovegetative profiles, different degrees of cognitive-emotional vulnerability and a higher or a lower level of acceptance of the illness could be supposed. Finally, recent findings defend the idea of the traumatic experiences as a determining factor to develop a SD.

In accordance to the last notions regarding the SD, some therapeutic approaches could be interesting specifically techniques focusing on the vagal nerve. In this context, biofeedback [BFB] could provide a powerful method to restore the clinical and physiological impairments.

As a consequence, the main objective is to evaluate the physiological and clinical effects of the BFB training with patients suffering from SD: Irritable Bowel Syndrome [IBS] or Psychogenic Non Epileptic Seizure [PNES]. The investigators make the prediction that the patients will be more or less responding to the biofeedback depending on their neurovegetative profile. A clustering will be performed in advance to identify the patients having a dysfunctional neurovegetative profile and patients having a functional neurovegetative profile. It will also permit to the investigators to confirm the hypothesis about the existence of two neurovegetative profiles related to a visceral-brain decoupling concerning the SD, independently of its form. To attest to it, 2 types of somatoform disorders will be analyzed: the irritable bowel syndrome manifesting by peripheral symptoms and the psychogenic non-epileptic seizures manifesting by central symptoms. Then the investigators will carry out a psycho-social exploration to demonstrate a higher cognitive-emotional vulnerability and a higher traumatic event incidence in this particular population, depending on their autonomic profiles.

ELIGIBILITY:
Inclusion Criteria:

* Somatoform disorders (IBS or PNES) diagnosis must be established by the partner doctors
* Participants must have home computer
* Participants must be of the age of majority
* Participants must be registered for social security
* Participants must have signed an informed consent

Exclusion Criteria:

* Specially protected participants (under clauses L1121-5 and L1121-8 by the code of public health): juveniles, pregnant womens, nursing mothers, law's protection peoples
* Participants suffering from a severe psychiatric disease needing specialised attention
* Participants suffering from or have suffered from a severe disease causing autonomic dysfunctions (heart failure, asthma, blood disease, renal failure, peripheral neuropathy, vagotomy, thyroid disorder, alcoholism, liver disease, amyloidosis)
* Participants taking medication which could be impact autonomic nervous system activity (anticholinergic, antiarrhythmics, clonidine, beta-blockers, tricyclic anti-depressants, metronidazole)
* Participants placing under judicial or administrative supervisions
* Participants were compensated more than 4500 euros because of his research protocol participation concerning human over the 12 months prior to the actual study
* Participants being not be able to contact in emergency
* Participants being in an exclusion period from another study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-09-05 (Actual)

PRIMARY OUTCOMES:
High frequency [HF] (0.15-0.40 Hz) | Day 1 (T1)
  High frequency (0.15-0.40 Hz), frequency-domain parameter
  HF will be measured using the electrocardiogram [ECG]:
  ECG data will be recorded using 3 single use and adhesive electrodes placed on the inner side of the right wrist, on the right shoulder and on the left side in accordance with the DII standard position (Einthoven). Physiological data recorded are related to the heart rate variability [HRV].
High frequency [HF] (0.15-0.40 Hz) | Up to 25 days from T1 (T2)
  High frequency (0.15-0.40 Hz), frequency-domain parameter
  HF will be measured using the electrocardiogram [ECG]:
  ECG data will be recorded using 3 single use and adhesive electrodes placed on the inner side of the right wrist, on the right shoulder and on the left side in accordance with the DII standard position (Einthoven). Physiological data recorded are related to the heart rate variability [HRV].
High frequency [HF] (0.15-0.40 Hz) | Up to 52 days from T1 (T3)
  High frequency (0.15-0.40 Hz), frequency-domain parameter
  HF will be measured using the electrocardiogram [ECG]:
  ECG data will be recorded using 3 single use and adhesive electrodes placed on the inner side of the right wrist, on the right shoulder and on the left side in accordance with the DII standard position (Einthoven). Physiological data recorded are related to the heart rate variability [HRV].
Root mean square of successive RR interval differences [RMSSD] | Day 1 (T1)
  Root mean square of successive RR interval differences, temporal-domain parameter
  RMSSD will be measured using the electrocardiogram [ECG]:
  ECG data will be recorded using 3 single use and adhesive electrodes placed on the inner side of the right wrist, on the right shoulder and on the left side in accordance with the DII standard position (Einthoven). Physiological data recorded are related to the heart rate variability [HRV].
Root mean square of successive RR interval differences [RMSSD] | Up to 25 days from T1 (T2)
  Root mean square of successive RR interval differences, temporal-domain parameter
  RMSSD will be measured using the electrocardiogram [ECG]:
  ECG data will be recorded using 3 single use and adhesive electrodes placed on the inner side of the right wrist, on the right shoulder and on the left side in accordance with the DII standard position (Einthoven). Physiological data recorded are related to the heart rate variability [HRV].
Root mean square of successive RR interval differences [RMSSD] | Up to 52 days from T1 (T3)
  Root mean square of successive RR interval differences, temporal-domain parameter
  RMSSD will be measured using the electrocardiogram [ECG]:
  ECG data will be recorded using 3 single use and adhesive electrodes placed on the inner side of the right wrist, on the right shoulder and on the left side in accordance with the DII standard position (Einthoven). Physiological data recorded are related to the heart rate variability [HRV].

SECONDARY OUTCOMES:
Low frequency [LF] (0.04-0.15 Hz) | Day 1 (T1)
  Low frequency (0.04-0.15 Hz), frequency-domain parameter
  LF will be measured using the electrocardiogram [ECG]:
  ECG data will be recorded using 3 single use and adhesive electrodes placed on the inner side of the right wrist, on the right shoulder and on the left side in accordance with the DII standard position (Einthoven). Physiological data recorded are related to the heart rate variability [HRV].
Low frequency [LF] (0.04-0.15 Hz) | Up to 25 days from T1 (T2)
  Low frequency (0.04-0.15 Hz), frequency-domain parameter
  LF will be measured using the electrocardiogram [ECG]:
  ECG data will be recorded using 3 single use and adhesive electrodes placed on the inner side of the right wrist, on the right shoulder and on the left side in accordance with the DII standard position (Einthoven). Physiological data recorded are related to the heart rate variability [HRV].
Low frequency [LF] (0.04-0.15 Hz) | Up to 52 days from T1 (T3)
  Low frequency (0.04-0.15 Hz), frequency-domain parameter
  LF will be measured using the electrocardiogram [ECG]:
  ECG data will be recorded using 3 single use and adhesive electrodes placed on the inner side of the right wrist, on the right shoulder and on the left side in accordance with the DII standard position (Einthoven). Physiological data recorded are related to the heart rate variability [HRV].
Low frequency [LF] 0.1 Hertz (0.075-0.108Hz) | Day 1 (T1)
  Spectral power of the low-frequency 0.1Hz band (0.075-0.108Hz), frequency-domain parameter
  LF-0.1Hz will be measured using the electrocardiogram [ECG]:
  ECG data will be recorded using 3 single use and adhesive electrodes placed on the inner side of the right wrist, on the right shoulder and on the left side in accordance with the DII standard position (Einthoven). Physiological data recorded are related to the heart rate variability [HRV].
Low frequency [LF] 0.1 Hertz (0.075-0.108Hz) | Up to 25 days from T1 (T2)
  Spectral power of the low-frequency 0.1Hz band (0.075-0.108Hz), frequency-domain parameter
  LF-0.1Hz will be measured using the electrocardiogram [ECG]:
  ECG data will be recorded using 3 single use and adhesive electrodes placed on the inner side of the right wrist, on the right shoulder and on the left side in accordance with the DII standard position (Einthoven). Physiological data recorded are related to the heart rate variability [HRV].
Low frequency [LF] 0.1 Hertz (0.075-0.108Hz) | Up to 52 days from T1 (T3)
  Spectral power of the low-frequency 0.1Hz band (0.075-0.108Hz), frequency-domain parameter
  LF-0.1Hz will be measured using the electrocardiogram [ECG]:
  ECG data will be recorded using 3 single use and adhesive electrodes placed on the inner side of the right wrist, on the right shoulder and on the left side in accordance with the DII standard position (Einthoven). Physiological data recorded are related to the heart rate variability [HRV].
Total power (0-0.40 Hz) | Day 1 (T1)
  Total power of the 0-0.40 Hertz band, frequency-domain parameter
  Total power will be measured using the electrocardiogram [ECG]:
  ECG data will be recorded using 3 single use and adhesive electrodes placed on the inner side of the right wrist, on the right shoulder and on the left side in accordance with the DII standard position (Einthoven). Physiological data recorded are related to the heart rate variability [HRV].
Total power (0-0.40 Hz) | Up to 25 days from T1 (T2)
  Total power of the 0-0.40 Hertz band, frequency-domain parameter
  Total power will be measured using the electrocardiogram [ECG]:
  ECG data will be recorded using 3 single use and adhesive electrodes placed on the inner side of the right wrist, on the right shoulder and on the left side in accordance with the DII standard position (Einthoven). Physiological data recorded are related to the heart rate variability [HRV].
Total power (0-0.40 Hz) | Up to 52 days from T1 (T3)
  Total power of the 0-0.40 Hertz band, frequency-domain parameter
  Total power will be measured using the electrocardiogram [ECG]:
  ECG data will be recorded using 3 single use and adhesive electrodes placed on the inner side of the right wrist, on the right shoulder and on the left side in accordance with the DII standard position (Einthoven). Physiological data recorded are related to the heart rate variability [HRV].
Ratio Low frequency / High frequency [LF / HF] | Day 1 (T1)
  Ratio of LF to HF power, frequency-domain parameter
  LF/HF will be measured using the electrocardiogram [ECG]:
  ECG data will be recorded using 3 single use and adhesive electrodes placed on the inner side of the right wrist, on the right shoulder and on the left side in accordance with the DII standard position (Einthoven). Physiological data recorded are related to the heart rate variability [HRV].
Ratio Low frequency / High frequency [LF / HF] | Up to 25 days from T1 (T2)
  Ratio of LF to HF power, frequency-domain parameter
  LF/HF will be measured using the electrocardiogram [ECG]:
  ECG data will be recorded using 3 single use and adhesive electrodes placed on the inner side of the right wrist, on the right shoulder and on the left side in accordance with the DII standard position (Einthoven). Physiological data recorded are related to the heart rate variability [HRV].
Ratio Low frequency / High frequency [LF / HF] | Up to 52 days from T1 (T3)
  Ratio of LF to HF power, frequency-domain parameter
  LF/HF will be measured using the electrocardiogram [ECG]:
  ECG data will be recorded using 3 single use and adhesive electrodes placed on the inner side of the right wrist, on the right shoulder and on the left side in accordance with the DII standard position (Einthoven). Physiological data recorded are related to the heart rate variability [HRV].
Standard deviation of all NN intervals [SDNN] | Day 1 (T1)
  Standard deviation of all NN intervals, temporal-domain parameter
  SDNN will be measured using the electrocardiogram [ECG]:
  ECG data will be recorded using 3 single use and adhesive electrodes placed on the inner side of the right wrist, on the right shoulder and on the left side in accordance with the DII standard position (Einthoven). Physiological data recorded are related to the heart rate variability [HRV].
Standard deviation of all NN intervals [SDNN] | Up to 25 days from T1 (T2)
  Standard deviation of all NN intervals, temporal-domain parameter
  SDNN will be measured using the electrocardiogram [ECG]:
  ECG data will be recorded using 3 single use and adhesive electrodes placed on the inner side of the right wrist, on the right shoulder and on the left side in accordance with the DII standard position (Einthoven). Physiological data recorded are related to the heart rate variability [HRV].
Standard deviation of all NN intervals [SDNN] | Up to 52 days from T1 (T3)
  Standard deviation of all NN intervals, temporal-domain parameter
  SDNN will be measured using the electrocardiogram [ECG]:
  ECG data will be recorded using 3 single use and adhesive electrodes placed on the inner side of the right wrist, on the right shoulder and on the left side in accordance with the DII standard position (Einthoven). Physiological data recorded are related to the heart rate variability [HRV].
Skin conductance responses [SCR] frequency | Day 1 (T1)
  Skin conductance responses [SCR] frequency : number of the spontaneous galvanic skin responses by periods
  SCR will be measured using the Galvanic skin responses [GSR]:
  GSR data will be recorded using 2 skin sensors placed on the third phalanx of the forefinger and of the middle finger of the left hand. Physiological data recorded are related to the cholinergic sympathetic activity (tonic GSR / phasic GSR).
Skin conductance responses [SCR] frequency | Up to 25 days from T1 (T2)
  Skin conductance responses [SCR] frequency : number of the spontaneous galvanic skin responses by periods
  SCR will be measured using the Galvanic skin responses [GSR]:
  GSR data will be recorded using 2 skin sensors placed on the third phalanx of the forefinger and of the middle finger of the left hand. Physiological data recorded are related to the cholinergic sympathetic activity (tonic GSR / phasic GSR).
Skin conductance responses [SCR] frequency | Up to 52 days from T1 (T3)
  Skin conductance responses [SCR] frequency : number of the spontaneous galvanic skin responses by periods
  SCR will be measured using the Galvanic skin responses [GSR]:
  GSR data will be recorded using 2 skin sensors placed on the third phalanx of the forefinger and of the middle finger of the left hand. Physiological data recorded are related to the cholinergic sympathetic activity (tonic GSR / phasic GSR).
Skin conductance responses [SCR] amplitude | Day 1 (T1)
  Skin conductance responses amplitude: amplitude of the spontaneous galvanic skin responses by periods
  SCR will be measured using the Galvanic skin responses [GSR]:
  GSR data will be recorded using 2 skin sensors placed on the third phalanx of the forefinger and of the middle finger of the left hand. Physiological data recorded are related to the cholinergic sympathetic activity (tonic GSR / phasic GSR).
Skin conductance responses [SCR] amplitude | Up to 25 days from T1 (T2)
  Skin conductance responses amplitude: amplitude of the spontaneous galvanic skin responses by periods
  SCR will be measured using the Galvanic skin responses [GSR]:
  GSR data will be recorded using 2 skin sensors placed on the third phalanx of the forefinger and of the middle finger of the left hand. Physiological data recorded are related to the cholinergic sympathetic activity (tonic GSR / phasic GSR).
Skin conductance responses [SCR] amplitude | Up to 52 days from T1 (T3)
  Skin conductance responses amplitude: amplitude of the spontaneous galvanic skin responses by periods
  SCR will be measured using the Galvanic skin responses [GSR]:
  GSR data will be recorded using 2 skin sensors placed on the third phalanx of the forefinger and of the middle finger of the left hand. Physiological data recorded are related to the cholinergic sympathetic activity (tonic GSR / phasic GSR).
Integrated skin conductance responses [ISCR] | Day 1 (T1)
  Integrated skin conductance responses [ISCR]: area of the galvanic skin responses identified on the signal
  ISCR will be measured using the Galvanic skin responses [GSR]:
  GSR data will be recorded using 2 skin sensors placed on the third phalanx of the forefinger and of the middle finger of the left hand. Physiological data recorded are related to the cholinergic sympathetic activity (tonic GSR / phasic GSR).
Integrated skin conductance responses [ISCR] | Up to 25 days from T1 (T2)
  Integrated skin conductance responses [ISCR]: area of the galvanic skin responses identified on the signal
  ISCR will be measured using the Galvanic skin responses [GSR]:
  GSR data will be recorded using 2 skin sensors placed on the third phalanx of the forefinger and of the middle finger of the left hand. Physiological data recorded are related to the cholinergic sympathetic activity (tonic GSR / phasic GSR).
Integrated skin conductance responses [ISCR] | Up to 52 days from T1 (T3)
  Integrated skin conductance responses [ISCR]: area of the galvanic skin responses identified on the signal
  ISCR will be measured using the Galvanic skin responses [GSR]:
  GSR data will be recorded using 2 skin sensors placed on the third phalanx of the forefinger and of the middle finger of the left hand. Physiological data recorded are related to the cholinergic sympathetic activity (tonic GSR / phasic GSR).
Pulsatility index variation [PI] | Day 1 (T1)
  Pulsatility index variation [PI] : transit time flow
  PI will be measured using the Photoplethysmography [PPG]:
  PPG data will be recorded using a finger sensor. Physiological data recorded are related to the adrenergic sympathetic tone and allowing a record of the blood pulse waves associated with the heart rate.
Pulsatility index variation [PI] | Up to 25 days from T1 (T2)
  Pulsatility index variation [PI] : transit time flow
  PI will be measured using the Photoplethysmography [PPG]:
  PPG data will be recorded using a finger sensor. Physiological data recorded are related to the adrenergic sympathetic tone and allowing a record of the blood pulse waves associated with the heart rate.
Pulsatility index variation [PI] | Up to 52 days from T1 (T3)
  Pulsatility index variation [PI] : transit time flow
  PI will be measured using the Photoplethysmography [PPG]:
  PPG data will be recorded using a finger sensor. Physiological data recorded are related to the adrenergic sympathetic tone and allowing a record of the blood pulse waves associated with the heart rate.
Breathing rate | Day 1 (T1)
  Breathing rate by cycles per minute
  The breathing rate will be measured using a breathing belt.
Breathing rate | Up to 25 days from T1 (T2)
  Breathing rate by cycles per minute
  The breathing rate will be measured using a breathing belt.
Breathing rate | Up to 52 days from T1 (T3)
  Breathing rate by cycles per minute
  The breathing rate will be measured using a breathing belt.
Dominant power (0-0.15Hz) | Day 1 (T1)
  Dominant power of the 0-0.15 Hertz band, frequency-domain parameter
  Dominant power will be measured using the electrogastrogram [EGG]:
  EGG data will be recorded using 6 single use and adhesive electrodes placed on the skin of the abdomen.
Dominant power (0-0.15Hz) | Up to 25 days from T1 (T2)
  Dominant power of the 0-0.15 Hertz band, frequency-domain parameter
  Dominant power will be measured using the electrogastrogram [EGG]:
  EGG data will be recorded using 6 single use and adhesive electrodes placed on the skin of the abdomen.
Dominant power (0-0.15Hz) | Up to 52 days from T1 (T3)
  Dominant power of the 0-0.15 Hertz band, frequency-domain parameter
  Dominant power will be measured using the electrogastrogram [EGG]:
  EGG data will be recorded using 6 single use and adhesive electrodes placed on the skin of the abdomen.
Total power (0-0.15Hz) | Day 1 (T1)
  Total power of the 0-0.15 Hertz band, frequency-domain parameter
  Total power will be measured using the electrogastrogram [EGG]:
  EGG data will be recorded using 6 single use and adhesive electrodes placed on the skin of the abdomen.
Total power (0-0.15Hz) | Up to 25 days from T1 (T2)
  Total power of the 0-0.15 Hertz band, frequency-domain parameter
  Total power will be measured using the electrogastrogram [EGG]:
  EGG data will be recorded using 6 single use and adhesive electrodes placed on the skin of the abdomen.
Total power (0-0.15Hz) | Up to 52 days from T1 (T3)
  Total power of the 0-0.15 Hertz band, frequency-domain parameter
  Total power will be measured using the electrogastrogram [EGG]:
  EGG data will be recorded using 6 single use and adhesive electrodes placed on the skin of the abdomen.
Slow-waves frequency (physiological outcome) | Day 1 (T1)
  Slow-waves frequency per minute, frequency-domain parameter
  Slow-wave frequency will be measured using the electrogastrogram [EGG]:
  EGG data will be recorded using 6 single use and adhesive electrodes placed on the skin of the abdomen.
Slow-waves frequency (physiological outcome) | Up to 25 days from T1 (T2)
  Slow-waves frequency per minute, frequency-domain parameter
  Slow-wave frequency will be measured using the electrogastrogram [EGG]:
  EGG data will be recorded using 6 single use and adhesive electrodes placed on the skin of the abdomen.
Slow-waves frequency (physiological outcome) | Up to 52 days from T1 (T3)
  Slow-waves frequency per minute, frequency-domain parameter
  Slow-wave frequency will be measured using the electrogastrogram [EGG]:
  EGG data will be recorded using 6 single use and adhesive electrodes placed on the skin of the abdomen.
Delta frequency (0-4Hz) | Day 1 (T1)
  Delta frequency 0-4 Hertz band
  Delta frequency will be measured using the electroencephalogram [EEG]:
  EEG data will be recorded using a EEG headsets including 64 electrodes. The EEG is related to the brain activity generated by the neural functioning.
Delta frequency (0-4Hz) | Up to 25 days from T1 (T2)
  Delta frequency 0-4 Hertz band
  Delta frequency will be measured using the electroencephalogram [EEG]:
  EEG data will be recorded using a EEG headsets including 64 electrodes. The EEG is related to the brain activity generated by the neural functioning.
Delta frequency (0-4Hz) | Up to 52 days from T1 (T3)
  Delta frequency 0-4 Hertz band
  Delta frequency will be measured using the electroencephalogram [EEG]:
  EEG data will be recorded using a EEG headsets including 64 electrodes. The EEG is related to the brain activity generated by the neural functioning.
Theta frequency (4-7Hz) | Day 1 (T1)
  Theta frequency 4-7 Hertz band
  Theta frequency will be measured using the electroencephalogram [EEG]:
  EEG data will be recorded using a EEG headsets including 64 electrodes. The EEG is related to the brain activity generated by the neural functioning.
Theta frequency (4-7Hz) | Up to 25 days from T1 (T2)
  Theta frequency 4-7 Hertz band
  Theta frequency will be measured using the electroencephalogram [EEG]:
  EEG data will be recorded using a EEG headsets including 64 electrodes. The EEG is related to the brain activity generated by the neural functioning.
Theta frequency (4-7Hz) | Up to 52 days from T1 (T3)
  Theta frequency 4-7 Hertz band
  Theta frequency will be measured using the electroencephalogram [EEG]:
  EEG data will be recorded using a EEG headsets including 64 electrodes. The EEG is related to the brain activity generated by the neural functioning.
Alpha frequency (8-12Hz) | Day 1 (T1)
  Alpha frequency 8-12 Hertz band
  Alpha frequency will be measured using the electroencephalogram [EEG]:
  EEG data will be recorded using a EEG headsets including 64 electrodes. The EEG is related to the brain activity generated by the neural functioning.
Alpha frequency (8-12Hz) | Up to 25 days from T1 (T2)
  Alpha frequency 8-12 Hertz band
  Alpha frequency will be measured using the electroencephalogram [EEG]:
  EEG data will be recorded using a EEG headsets including 64 electrodes. The EEG is related to the brain activity generated by the neural functioning.
Alpha frequency (8-12Hz) | Up to 52 days from T1 (T3)
  Alpha frequency 8-12 Hertz band
  Alpha frequency will be measured using the electroencephalogram [EEG]:
  EEG data will be recorded using a EEG headsets including 64 electrodes. The EEG is related to the brain activity generated by the neural functioning.
Beta frequency (13-30Hz) | Day 1 (T1)
  Beta frequency 13-30 Hertz band
  Beta frequency will be measured using the electroencephalogram [EEG]:
  EEG data will be recorded using a EEG headsets including 64 electrodes. The EEG is related to the brain activity generated by the neural functioning.
Beta frequency (13-30Hz) | Up to 25 days from T1 (T2)
  Beta frequency 13-30 Hertz band
  Beta frequency will be measured using the electroencephalogram [EEG]:
  EEG data will be recorded using a EEG headsets including 64 electrodes. The EEG is related to the brain activity generated by the neural functioning.
Beta frequency (13-30Hz) | Up to 52 days from T1 (T3)
  Beta frequency 13-30 Hertz band
  Beta frequency will be measured using the electroencephalogram [EEG]:
  EEG data will be recorded using a EEG headsets including 64 electrodes. The EEG is related to the brain activity generated by the neural functioning.
Gamma frequency (>30Hz) | Day 1 (T1)
  Gamma frequency >30 Hertz band
  Gamma frequency will be measured using the electroencephalogram [EEG]:
  EEG data will be recorded using a EEG headsets including 64 electrodes. The EEG is related to the brain activity generated by the neural functioning.
Gamma frequency (>30Hz) | Up to 25 days from T1 (T2)
  Gamma frequency >30 Hertz band
  Gamma frequency will be measured using the electroencephalogram [EEG]:
  EEG data will be recorded using a EEG headsets including 64 electrodes. The EEG is related to the brain activity generated by the neural functioning.
Gamma frequency (>30Hz) | Up to 52 days from T1 (T3)
  Gamma frequency >30 Hertz band
  Gamma frequency will be measured using the electroencephalogram [EEG]:
  EEG data will be recorded using a EEG headsets including 64 electrodes. The EEG is related to the brain activity generated by the neural functioning.
Alexithymia score | Up to 16 days from T2
  Alexithymia score will be measured using the Bermond-Vorst Alexithymia Questionnaire B version (BVAQ-B; Vorst & Bermond, 2001; French version Deborde et al., 2004). The subscale as considered as a trait scale including 20 items.
Neuroticism score | Up to 16 days from T1
  Neuroticism score will be measured using the Big Five Inventory-Neuroticism (BFI-N; John et al., 1991; French version Plaisant et al., 2005). The subscale as considered as a trait scale including 8 items.
Trait and state anxiety scores | Up to 8 days from T1
  The trai and state anxiety scores will be measured using the State-Trait Anxiety Inventory (STAI Y-AB) (Spielberger et al., 1983; French version Bruchon-Schweitzer & Paulhan, 1990). The scale includes 40 items.
Style of coping | Up to 16 days from T1
  The style of coping will be measured using the Brief Cope (Carver, 1997; French version Muller & Spitz, 2003). We will use it in its trait version. The subscale as considered as a trait scale including 28 items.
Positive affectivity score | Day 1 (T1)
  Positive affectivity score will be measured using the Positive And Negative Affect Schedule (PANAS; Watson et al., 1988; French version Caci & Bayle, 2007). To measure a global affective state, a score of positivity will be calculated by subtracting negative affect score from positive affect score. The subscale as considered as a state scale including 20 items.
Positive affectivity score | Up to 25 days from T1 (T2)
  Positive affectivity score will be measured using the Positive And Negative Affect Schedule (PANAS; Watson et al., 1988; French version Caci & Bayle, 2007). To measure a global affective state, a score of positivity will be calculated by subtracting negative affect score from positive affect score. The subscale as considered as a state scale including 20 items.
Positive affectivity score | Up to 52 days from T1 (T3)
  Positive affectivity score will be measured using the Positive And Negative Affect Schedule (PANAS; Watson et al., 1988; French version Caci & Bayle, 2007). To measure a global affective state, a score of positivity will be calculated by subtracting negative affect score from positive affect score. The subscale as considered as a state scale including 20 items.
Depressive symptoms score | Day 1 (T1)
  The depressive symptoms score will be measured using the Center for Epidemiologic Studies-Depression Scale (CES-D; Radloff, 1977; French version Führer & Rouillon, 1989). The subscale as considered as a state scale including 20 items.
Depressive symptoms score | Up to 25 days from T1 (T2)
  The depressive symptoms score will be measured using the Center for Epidemiologic Studies-Depression Scale (CES-D; Radloff, 1977; French version Führer & Rouillon, 1989). The subscale as considered as a state scale including 20 items.
Depressive symptoms score | Up to 52 days from T1 (T3)
  The depressive symptoms score will be measured using the Center for Epidemiologic Studies-Depression Scale (CES-D; Radloff, 1977; French version Führer & Rouillon, 1989). The subscale as considered as a state scale including 20 items.
Perceived-stress level | Day 1 (T1)
  The perceived-stress level will be measured using the Perceived Stress Scale (PSS; Cohen et al., 1983; French version Bellighausen et al., 2009). The subscale as considered as a state scale including 10 items.
Perceived-stress level | Up to 25 days from T1 (T2)
  The perceived-stress level will be measured using the Perceived Stress Scale (PSS; Cohen et al., 1983; French version Bellighausen et al., 2009). The subscale as considered as a state scale including 10 items.
Perceived-stress level | Up to 52 days from T1 (T3)
  The perceived-stress level will be measured using the Perceived Stress Scale (PSS; Cohen et al., 1983; French version Bellighausen et al., 2009). The subscale as considered as a state scale including 10 items.
Coping flexibility | Day 1 (T1)
  The coping flexibility score will be measured using the Coping Flexibility Scale (CFS; Kato, 2012). The CFS measures the coping flexibility including 10 items. The subscale as considered as a state scale.
Coping flexibility | Up to 25 days from T1 (T2)
  The coping flexibility score will be measured using the Coping Flexibility Scale (CFS; Kato, 2012). The CFS measures the coping flexibility including 10 items. The subscale as considered as a state scale.
Coping flexibility | Up to 52 days from T1 (T3)
  The coping flexibility score will be measured using the Coping Flexibility Scale (CFS; Kato, 2012). The CFS measures the coping flexibility including 10 items. The subscale as considered as a state scale.
Metacoping | Day 1 (T1)
  The metacoping score will be measured using a visual analogue scale (VAS). The VAS was developed by ourselves to measure the perceived effectiveness of coping by asking: " how strategies used by yourself to cope with the situation were efficient? ". The participants will have to rate from 0 (no efficacy) to 10 (maximum of efficacy). The subscale as considered as a state scale.
Metacoping | Up to 25 days from T1 (T2)
  The metacoping score will be measured using a visual analogue scale (VAS). The VAS was developed by ourselves to measure the perceived effectiveness of coping by asking: " how strategies used by yourself to cope with the situation were efficient? ". The participants will have to rate from 0 (no efficacy) to 10 (maximum of efficacy). The subscale as considered as a state scale.
Metacoping | Up to 52 days from T1 (T3)
  The metacoping score will be measured using a visual analogue scale (VAS). The VAS was developed by ourselves to measure the perceived effectiveness of coping by asking: " how strategies used by yourself to cope with the situation were efficient? ". The participants will have to rate from 0 (no efficacy) to 10 (maximum of efficacy). The subscale as considered as a state scale.
Social support score | Up to 8 days from T1
  The social support score will be measured using the Social Support Questionnaire short version (SSQ6; Sarason et al., 1987a; French version Bruchon-Schweitzer et al., 2003). The subscale as considered as a trait scale including 6 items.
Interceptive sensitivity score | Up to 8 days from T1
  The interceptive sensitivity score will be measured using the Multidimensional Assessment of Interoceptive Awareness second version (MAIA-2; Mehling et al., 2018). The subscale as considered as a trait scale including 37 items.
Life satisfaction score | Day 1 (T1)
  The life satisfaction score will be measured using the Satisfaction With Life Scale (SWLS; Diener et al., 1985; French version Blais et al., 1989). The subscale as considered as a state scale including 5 items.
Life satisfaction score | Up to 25 days from T1 (T2)
  The life satisfaction score will be measured using the Satisfaction With Life Scale (SWLS; Diener et al., 1985; French version Blais et al., 1989). The subscale as considered as a state scale including 5 items.
Life satisfaction score | Up to 52 days from T1 (T3)
  The life satisfaction score will be measured using the Satisfaction With Life Scale (SWLS; Diener et al., 1985; French version Blais et al., 1989). The subscale as considered as a state scale including 5 items.
Negative impact scores | Up to 16 days from T2
  The negative impact score will be measured using the Life Experiences Survey (LES; Sarason et al., 1978). The subscale as considered as a trait scale including 50 items. In this study a modified version of the LES will be used, whereby subjects documented the presence and perceived impact of adulthood life events that had occurred since 18 years of age to the time of completion of the survey. For the purposes of this study, 3 scores will be generated from this survey: the number of negatively perceived life events, the negative impact score determined by the sum of the impact scores of negatively perceived life events alone (higher scores indicate greater negative impact), and the total impact score determined by the sum of the impact scores of both negatively and positively perceived life events (higher scores indicate an overall more positive impact and lower scores indicate an overall more negative impact of all adulthood life events).
Frequency, severity and intensity scores | Up to 8 days from T2
  The frequency, severity and intensity scores will be measured using the Daily Hassles Scale (DHS; Kanner et al., 1981). The subscale as considered as a trait scale including 117 items.
Child Abuse scores | Up to 16 days from T1
  The child abuse scores will be measured using the Childhood Trauma Questionnaire-Short Form (CTQ; Bernstein et al., 2003). The subscale as considered as a trait scale including 28 items.
Acceptance score | Day 1 (T1)
  The acceptance score will be measured using the Illness Cognition Questionnaire for chronic disease (ICQ-18; Evers et al., 2001). The subscale as considered as a state scale including 18 items.
Acceptance score | Up to 25 days from T1 (T2)
  The acceptance score will be measured using the Illness Cognition Questionnaire for chronic disease (ICQ-18; Evers et al., 2001). The subscale as considered as a state scale including 18 items.
Acceptance score | Up to 52 days from T1 (T3)
  The acceptance score will be measured using the Illness Cognition Questionnaire for chronic disease (ICQ-18; Evers et al., 2001). The subscale as considered as a state scale including 18 items.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno BONAZ, Pr, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital, Grenoble Alpes, Grenoble, Isère, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Laborde S, Mosley E, Thayer JF. Heart Rate Variability and Cardiac Vagal Tone in Psychophysiological Research - Recommendations for Experiment Planning, Data Analysis, and Data Reporting. Front Psychol. 2017 Feb 20;8:213. doi: 10.3389/fpsyg.2017.00213. eCollection 2017. PMID 28265249
- [Background] Muller L, Spitz E. [Multidimensional assessment of coping: validation of the Brief COPE among French population]. Encephale. 2003 Nov-Dec;29(6):507-18. French. PMID 15029085
- [Background] Mehling WE, Acree M, Stewart A, Silas J, Jones A. The Multidimensional Assessment of Interoceptive Awareness, Version 2 (MAIA-2). PLoS One. 2018 Dec 4;13(12):e0208034. doi: 10.1371/journal.pone.0208034. eCollection 2018. PMID 30513087
- [Background] Varon C, Morales J, Lazaro J, Orini M, Deviaene M, Kontaxis S, Testelmans D, Buyse B, Borzee P, Sornmo L, Laguna P, Gil E, Bailon R. A Comparative Study of ECG-derived Respiration in Ambulatory Monitoring using the Single-lead ECG. Sci Rep. 2020 Mar 31;10(1):5704. doi: 10.1038/s41598-020-62624-5. PMID 32235865
- [Background] de Vroege L, Emons WHM, Sijtsma K, van der Feltz-Cornelis CM. Psychometric Properties of the Bermond-Vorst Alexithymia Questionnaire (BVAQ) in the General Population and a Clinical Population. Front Psychiatry. 2018 Apr 23;9:111. doi: 10.3389/fpsyt.2018.00111. eCollection 2018. PMID 29740350
- [Background] Bulut NS, Wurz A, Yorguner Kupeli N, Carkaxhiu Bulut G, Sungur MZ. Heart rate variability response to affective pictures processed in and outside of conscious awareness: Three consecutive studies on emotional regulation. Int J Psychophysiol. 2018 Jul;129:18-30. doi: 10.1016/j.ijpsycho.2018.05.006. Epub 2018 May 19. PMID 29787784
- [Background] Schumann A, Kohler S, Brotte L, Bar KJ. Effect of an eight-week smartphone-guided HRV-biofeedback intervention on autonomic function and impulsivity in healthy controls. Physiol Meas. 2019 Jul 1;40(6):064001. doi: 10.1088/1361-6579/ab2065. PMID 31071705
- [Background] Sarason IG, Johnson JH, Siegel JM. Assessing the impact of life changes: development of the Life Experiences Survey. J Consult Clin Psychol. 1978 Oct;46(5):932-46. doi: 10.1037//0022-006x.46.5.932. No abstract available. PMID 701572
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- See also: Vorst, Harrie C.M, et Bob Bermond. " Validity and Reliability of the Bermond-Vorst Alexithymia Questionnaire ". Personality and Individual Differences 30, no 3 (février 2001): 413 34. — https://doi.org/10.1016/S0191-8869(00)00033-7
- See also: Plaisant O, Srivastava S, Mendelsohn GA, Debray Q, John OP. Relations entre le Big Five Inventory franc¸ais et le manuel diagnostique des troubles mentaux dans un échantillon clinique franc¸ais. Ann Med Psychol 2005;163:161-7. — https://doi.org/10.1016/j.amp.2005.02.002
- See also: Radloff LS. The CES-D scale: a self report depression scalefor research in the general population. App Psycho Meas1977;1:384-401. — https://conservancy.umn.edu/items/38cff7f5-eb7a-4578-9a45-483e0bf5e697
- See also: Spielberger, C. D., Gorsuch, R. L., Luschene, R. E., Vagg, P. R., & Jacobs, G. A. (1983). Manual for the state-trait anxiety inventory form Y. CA: Mind Garden Press. — https://www.researchgate.net/publication/235361542_Manual_for_the_State-Trait_Anxiety_Inventory_Form_Y1_-_Y2

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-10): https://cdn.clinicaltrials.gov/large-docs/33/NCT04807933/Prot_SAP_000.pdf